CLINICAL TRIAL: NCT05043662
Title: A Prospective, Single-blinded Study of UroCAD Assay Combined With Computed Tomography Urography and Urine Cytology for UTUC Diagnosis.
Brief Title: UroCAD Assay Combined With Computed Tomography Urography and Urine Cytology for UTUC Diagnosis.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Shuxiong Zeng, M.D., Ph.D, Changhai Hospital
Other Study IDs: UroCAD-UTUC
Record Dates: First submitted 2021-09-05; First posted 2021-09-14 (Actual); Last update posted 2021-09-14 (Actual); Status verified 2021-09

CONDITIONS: Urothelial Carcinoma; Diagnoses Disease; Ureter Cancer; IMAGE; Cytology
Keywords: UTUC; CIN; cytology; CTU
MeSH Terms: conditions — Carcinoma, Transitional Cell; Ureteral Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The extracted DNA from morning urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Urothelial carcinoma group: The extracted DNA from morning urine will be analyzed by UroCAD to determine the level of CNV. CTU and cytology will be performed according to the routine of clinical practice (N=80).
  Interventions: Diagnostic Test: UroCAD assay, CTU examination and urine cytology
- Control group: Patients need to undergo CTU examination and being treated for benign diseases with ureteroscopy, but without any tumor will provide a negative control to provide data for determining the sensitivity and specificity of UroCAD, CTU and cytology assay (N=30).
  Interventions: Diagnostic Test: UroCAD assay, CTU examination and urine cytology

INTERVENTIONS:
Diagnostic Test: UroCAD assay, CTU examination and urine cytology — The extracted DNA from morning urine will be analyzed by UroCAD to determine the level of CNV. CTU and cytology will be performed according to the routine of clinical practice.

SUMMARY:
Upper tract urothelial carcinoma (UTUC) diagnosis include urography using computed tomography urography (CTU) or urography using MRI (MRU). The sensitivity of CTU decreases substan¬tially with decreasing lesion size. Other drawbacks of CTU include the radiation exposure and potential adverse effects in patients with allergic reactions or pre-existing renal impairment. In terms of urine cytology, the major drawbacks of urine cytology are low sensitivity and highly dependent of the experience and skills of the cytopathologist. We here intended to investigate whether UroCAD can be added in the diagnostic work-up of UTUC patient, and improve the accuracy of predicting UTUC before surgery.

DETAILED DESCRIPTION:
The recommendations for imaging in UTUC diagnosis include urography using CTU or MRU. In the standard diag¬nostic work up, urine cytology and a cystoscopy to rule out a concomitant bladder tumor are also advised. In addition, diagnostic ureterorenoscopy and biopsy are advised in patients in whom the findings of these pro¬cedures could influence treatment decisions, The sensitivity of CTU decreases substan¬tially with decreasing lesion size. For polypoid tumors of 5-10 mm maximal diameter, CTU has a high sensitivity and specificity, but sensitivity decreases to 89% for lesions <5 mm and further to 40% for lesions <3 mm. Flat lesions are even more difficult to diagnose. Other drawbacks of CTU include the radiation exposure and the need for intravenous contrast media with accompa¬nying potential adverse effects in patients with allergic reactions or pre-existing renal impairment. In terms of urine cytology, the major drawbacks of urine cytology tests: the sensitivity of positive urine cytology is highly dependent on tumor grade and decreases to 12% for low-grade tumors and 15% for non-invasive stage Ta tumors. Hence, low-grade urothelial tumors cannot be reliably detected by urine cytology. Finally, the accuracy of the cytology findings is highly dependent of the experience and skills of the cytopathologist. Our previous study has proved that UroCAD, which is able to detect chromosomal aberrations of the urine exfoliated cells, is a reliable method in diagnosing urothelial carcinoma with sensitivity and specificity of 82.5% and 96.9%, respectively. But its potential role in diagnosis of UTUC in combination with CTU and cytology hasn't been assessed yet and the accuracy of UroCAD in detecting UTUC still need to be further validated. We here intended to investigate whether UroCAD can be added in the diagnostic work-up of UTUC patient, and improve the accuracy of predicting UTUC before surgery.

ELIGIBILITY:
Inclusion Criteria:

Patients suspected with UTUC and planned to undergo surgery such as such ureteroscopy or radical nephroureterectomy.

Participants without any tumor disease and willing to attend the study by providing morning urine.

Male or female patients aged >= 18 years. Participants signed informed consent form.

Exclusion Criteria:

Individuals unwilling to sign the consent form or unwilling to provide morning urine for test or unwilling to provide the medical record.

Patient already received suprapubic cystostomy or urethral catheterization. Participants with late-stage uremia and need regular dialysis. Participants with reasons like elevated serum creatinine, allergy to intravenous CT contrast media et al, and unable to undergo CTU.

Patient with cancer other than urothelial carcinoma.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients suspected of UTUC or participants in control group from September 2021 to October 2022 in Changhai hospital
Sampling Method: Non-Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-10-01 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and Specificity of urinalysis by UroCAD assay combined with CTU and cytology | Through study completion, an average of 30 months
  Number of patients "declared positive" with the UroCAD assay, CTU or cytology among the patients suffered from UTUC and number of patients "declared negative" with these tests among the patients without cancer.

SECONDARY OUTCOMES:
Identification of the correlation between the level of CNV and the grade of the tumor sample | Through study completion, an average of 30 months
  Level of CNV in the urine sample compared with the grade of the tumor confirmed by histopathologic examination
Identification of the correlation between the level of CNV and the stage of the tumor sample | Through study completion, an average of 30 months
  Level of CNV in the urine sample compared with the stage of the tumor confirmed by histopathologic examination
Comparison of the sensitivity and specificity of the UroCAD analysis versus urine cytology and CTU | Through study completion, an average of 30 months
  Number of patients "declared positive" with the UroCAD analysis versus patients "declared positive" with the urine cytology or CTU, and number of patients "declared negative" with the UroCAD analysis versus patients " declared negative " with the urine cytology or CTU.

CONTACTS AND LOCATIONS:
Overall Officials: Chuangliang Xu, M.D., Ph.D, Study Director — Changhai Hospital
Locations (1):
- Changhai Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No
To pretect the personal privacy of participants and the genetic sequencing information, IPD data will not be shared.

REFERENCES:
- [Background] Baard J, de Bruin DM, Zondervan PJ, Kamphuis G, de la Rosette J, Laguna MP. Diagnostic dilemmas in patients with upper tract urothelial carcinoma. Nat Rev Urol. 2017 Mar;14(3):181-191. doi: 10.1038/nrurol.2016.252. Epub 2016 Dec 13. PMID 27958391
- [Background] Janisch F, Shariat SF, Baltzer P, Fajkovic H, Kimura S, Iwata T, Korn P, Yang L, Glybochko PV, Rink M, Abufaraj M. Diagnostic performance of multidetector computed tomographic (MDCTU) in upper tract urothelial carcinoma (UTUC): a systematic review and meta-analysis. World J Urol. 2020 May;38(5):1165-1175. doi: 10.1007/s00345-019-02875-8. Epub 2019 Jul 18. PMID 31321509
- [Result] Zeng S, Ying Y, Xing N, Wang B, Qian Z, Zhou Z, Zhang Z, Xu W, Wang H, Dai L, Gao L, Zhou T, Ji J, Xu C. Noninvasive Detection of Urothelial Carcinoma by Cost-effective Low-coverage Whole-genome Sequencing from Urine-Exfoliated Cell DNA. Clin Cancer Res. 2020 Nov 1;26(21):5646-5654. doi: 10.1158/1078-0432.CCR-20-0401. Epub 2020 Oct 9. PMID 33037018